CLINICAL TRIAL: NCT03459365
Title: A Prospective Pilot Study to Evaluate Efficacy and Safety of Euflexxa for the Treatment of Osteoarthritis
Brief Title: Euflexxa for the Treatment of Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Carlos Higuera-Rueda, Vice Chair for Quality and Patient Safety, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-1668
Record Dates: First submitted 2018-01-18; First posted 2018-03-08 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Euflexxa (Experimental): Two sets of Euflexxa injection at 0 and 6 months. Each set consists of 3 injections 1 week apart.
  Interventions: Device: Euflexxa

INTERVENTIONS:
Device: Euflexxa — Aspirations performed before each injection and at six weeks.

SUMMARY:
The effect of Euflexxa therapy for knee osteoarthritis on levels of inflammatory and degenerative synovial fluid bio-markers in patients with knee osteoarthritis

DETAILED DESCRIPTION:
The FLEXX trial was the first well-controlled, randomized, double-blind, multicenter study evaluating the efficacy of Euflexxa (1% sodium hyaluronate) therapy for knee osteoarthritis. Five-hundred-and-eighty patients were randomized to receive either Euflexxa or normal saline. There were significant improvements in the Visual analogue scale score Osteoarthritis Research Society International responder index, HRQoL, and function at 26-week follow-up.1 However, the FLEXX trial did not evaluate changes in synovial fluid bio-marker levels. The present study will be a prospective pilot study of 30 knees from subjects who receive intra-articular Euflexxa. The primary objective of this study is to prospectively determine, at 6-weeks, and 6-months post treatment, the changes in levels of synovial fluid biomarkers from pre- to post-injection in patients who receive Euflexxa. In addition, we will assess patient reported pain and patient reported outcomes up to 2 years from initiation of study.

ELIGIBILITY:
Inclusion criteria:

1. OA of the knee by American College of Rheumatology criteria
2. Those who failed non-pharmacological measures or simple analgesics
3. moderate to severe pain score of 41 to 90 mm recorded on 100-mm visual analog scale (VAS) immediately following a 50-foot walk
4. bilateral standing anterior-posterior radiograph demonstrating Kellgren and Lawrence grade 2 or 3 OA of the target knee
5. ability and willingness to use only acetaminophen as the analgesic (rescue) study medication
6. unassisted walking 50 feet on a flat surface and going up and down stairs
7. willingness and ability to complete efficacy and safety questionnaires

Exclusion criteria:

1. Age less than 18 years
2. any major injury to the target knee within the prior 12 months
3. any surgery to the target knee within the prior 12 months
4. surgery to the contralateral knee or other weight-bearing
5. inflammatory arthropathies
6. gout or pseudogout within the previous 6 months
7. radiographic acute fracture, severe loss of bone density, avascular necrosis, and/or severe bone or joint deformity in the target knee
8. osteonecrosis of either knee
9. fibromyalgia, pes anserine bursitis, lumbar radiculopathy, and/or neurogenic or vascular claudication
10. target knee joint infection or skin disorder/ infection within the previous 6 months
11. symptomatic OA of the hips, spine, or ankle; known hypersensitivity to acetaminophen, IA-BioHA, or phosphate-buffered saline solution
12. Women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the study
13. history of immune disorders; vascular insufficiency of lower limbs or peripheral neuropathy
14. current treatment or treatment of cancer within the previous 2 years (excluding basal cell or squamous cell carcinoma of the skin)
15. active liver or renal disease
16. any clinically significant abnormal laboratory value [to be defined in detail at a later point]
17. any intercurrent chronic disease or condition that might interfere with the completion of the study
18. participation in any experimental device study within the prior 6 months or any experimental drug study within the prior month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Higuera, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 30 knees (from 24 patients) recruited (some patients treated on both knees).
  7 knees withdrew from the study. 8 knees had dry taps. This left 15 knees from 11 patients with adequate baseline aspirates. One of the 1-month aspirates was too bloody to process, leaving 14 knees from 10 patients with adequate baseline and 1 month samples.
  3 knees had dry taps at 6 months, leaving 11 knees from 10 patients with adequate baseline, 1 month, and 6 month aspirates for data analysis.
Units Other Than Participants: Knees
Period: Overall Study
Arm/Group | Euflexxa
Started | 24; 30 Knees (30 knees from 24 patients enrolled)
Completed | 10; 11 Knees (11 knees from 10 patients)
Not Completed | 14; 19 Knees
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 8

BASELINE CHARACTERISTICS:
Population: 10 patients (11 knees). Baseline description is at the patient level (n=10)
Arm/Group | Euflexxa
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index, continuous [Mean (Standard Deviation); unit: kg/m^2] | 30 (7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hyaluronate Concentration
Description: The concentration of hyaluronate in the synovial fluid will be measured using Fluorophore-assisted carbohydrate electrophoresis. The difference between the mean concentration at baseline and 6 months is reported.
Time Frame: Baseline to 6 months
Population: 11 knees from 10 patients
Measure: Mean (Standard Deviation); unit: mg/ml
Units Other Than Participants: knees
Arm/Group | Euflexxa
Number analyzed (Participants) | 10
Number analyzed (knees) | 11
mg/ml | 0.29568 (1.65476)

2. Secondary Outcome: Changes in Tumor Necrosis Factor-stimulated Gene 6 (TSG-6)
Description: The levels of TSG-6 in the synovial fluid will be measured using Enzyme-linked immunosorbent assay. The difference in mean concentration between baseline and 6 months post injection is reported.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Units Other Than Participants: knees
Arm/Group | Euflexxa
Number analyzed (Participants) | 10
Number analyzed (knees) | 11
ng/ml | 3450 (5831)

3. Secondary Outcome: VAS Pain Score Improvement
Description: Change in VAS (visual analogue scale) pain score compared to baseline in the study cohort. VAS is a measure of pain with 0 being best and 10 being worst pain on a 10 cm scale (100 mm).
Time Frame: Baseline to 6 months
Population: 11 knees (10 patients)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: knees
Arm/Group | Euflexxa
Number analyzed (Participants) | 10
Number analyzed (knees) | 11
mm | 40 (13)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Euflexxa
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Euflexxa (N=10)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unrelated to the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT03459365/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03459365/ICF_001.pdf